CLINICAL TRIAL: NCT01030991
Title: Etiologic, Pathophysiologic, and Genetic Classification of Heart Failure With Preserved Ejection Fraction
Brief Title: Classification of Heart Failure With Preserved Ejection Fraction
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Sanjiv Shah, Associate Professor of Medicine, Northwestern University
Other Study IDs: AHA 0835488N
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Diastolic Heart Failure
Keywords: Heart failure; Ejection fraction; Diastolic heart failure; Diastolic dysfunction; Ventricular-arterial coupling; Exercise testing; Echocardiography; Tissue Doppler imaging; Arterial tonometry; Genetics; Epidemiology
MeSH Terms: conditions — Heart Failure, Diastolic; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Whole blood, saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HFpEF: HFpEF cohort (observational study)

SUMMARY:
The purpose of this study is to create a classification system for the heterogenous disorder of heart failure with preserved ejection fraction (HFpEF).

DETAILED DESCRIPTION:
Patients with HFpEF are a heterogeneous group with varying etiology and pathophysiology, which may play a large role in the difficulty in managing these patients and enrolling them in clinical trials. A major advance in the care of patients with HFpEF would be a classification system based on etiology, pathophysiology, and/or genetic factors as well as machine learning analyses. The ultimate goal of this study is to demonstrate that it is possible to better classify patients with HFpEF based on etiologic, pathophysiologic, and genetic differences between patients. If successful, this study could lead to: (1) novel risk estimation in patients with HFpEF and (2) more fruitful clinical trials based on targeting specific subsets of HFpEF.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years
* Signs or symptoms of congestive heart failure
* Left ventricular ejection fraction > 50%

Exclusion Criteria:

* Severe valvular heart disease
* History of cardiac transplantation
* Prior history of heart failure associated with left ventricular ejection fraction < 35%

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with signs or symptoms of heart failure with left ventricular ejection fraction > 50% are eligible for the study
Sampling Method: Non-Probability Sample
Enrollment: 514 (Actual)
Dates: Start 2008-07-01 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-05-21 (Actual)

PRIMARY OUTCOMES:
Heart failure hospitalization | 1 year
Cardiovascular hospitalization | 1 year
Mortality - all cause and cardiovascular | 1 year

SECONDARY OUTCOMES:
Exercise capacity (peak VO2) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv J Shah, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shah SJ, Katz DH, Selvaraj S, Burke MA, Yancy CW, Gheorghiade M, Bonow RO, Huang CC, Deo RC. Phenomapping for novel classification of heart failure with preserved ejection fraction. Circulation. 2015 Jan 20;131(3):269-79. doi: 10.1161/CIRCULATIONAHA.114.010637. Epub 2014 Nov 14. PMID 25398313
- [Derived] Rich JD, Burns J, Freed BH, Maurer MS, Burkhoff D, Shah SJ. Meta-Analysis Global Group in Chronic (MAGGIC) Heart Failure Risk Score: Validation of a Simple Tool for the Prediction of Morbidity and Mortality in Heart Failure With Preserved Ejection Fraction. J Am Heart Assoc. 2018 Oct 16;7(20):e009594. doi: 10.1161/JAHA.118.009594. PMID 30371285
- [Derived] Freed BH, Daruwalla V, Cheng JY, Aguilar FG, Beussink L, Choi A, Klein DA, Dixon D, Baldridge A, Rasmussen-Torvik LJ, Maganti K, Shah SJ. Prognostic Utility and Clinical Significance of Cardiac Mechanics in Heart Failure With Preserved Ejection Fraction: Importance of Left Atrial Strain. Circ Cardiovasc Imaging. 2016 Mar;9(3):10.1161/CIRCIMAGING.115.003754 e003754. doi: 10.1161/CIRCIMAGING.115.003754. PMID 26941415
- [Derived] Unger ED, Dubin RF, Deo R, Daruwalla V, Friedman JL, Medina C, Beussink L, Freed BH, Shah SJ. Association of chronic kidney disease with abnormal cardiac mechanics and adverse outcomes in patients with heart failure and preserved ejection fraction. Eur J Heart Fail. 2016 Jan;18(1):103-12. doi: 10.1002/ejhf.445. Epub 2015 Dec 3. PMID 26635076
- [Derived] Katz DH, Burns JA, Aguilar FG, Beussink L, Shah SJ. Albuminuria is independently associated with cardiac remodeling, abnormal right and left ventricular function, and worse outcomes in heart failure with preserved ejection fraction. JACC Heart Fail. 2014 Dec;2(6):586-96. doi: 10.1016/j.jchf.2014.05.016. Epub 2014 Oct 1. PMID 25282032
- See also: Northwestern University Heart Failure with Preserved Ejection Fraction (HFpEF) Program — http://www.hfpef.org